CLINICAL TRIAL: NCT07156864
Title: "Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of the Drug B10-FC - Study Drug for Early Etiotropic Therapy of Coronavirus Infection Caused by the SARS-CoV-2 Virus, Using Heavy-chain Humanized Monoclonal Antibodies, After Single Administration to Adult Patients".
Brief Title: "Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of the Drug B10-FC After Single Administration to Adult Patients".
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01-B5/В10-FC-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1/10 therapeutic dose (Experimental): 5 healthy volunteers + 1 healthy replacement volunteer will recieve 1/10 therapeutic dose of the study drug.
  Interventions: Drug: 1/10 therapeutic dose
- 1/2 therapeutic dose (Experimental): 5 healthy volunteers + 1 healthy replacement volunteer will recieve 1/2 therapeutic dose of the study drug.
  Interventions: Drug: 1/2 therapeutic dose
- full therapeutic dose (Experimental): 15 healthy volunteers + 3 healthy replacement volunteers will recieve full therapeutic dose of the study drug.
  Interventions: Drug: Patients with a verified diagnosis of COVID-19
- Patients with a verified diagnosis of COVID-19 (Experimental): 10 volunteers with a verified diagnosis of COVID-19 will recieve full therapeutic dose of the study drug.
  Interventions: Drug: full therapeutic dose

INTERVENTIONS:
Drug: 1/10 therapeutic dose — 5 volunteers + 1 replacement volunteer will recieve 1/10 therapeutic dose of the study drug (parenteral administration).
  Arms: 1/10 therapeutic dose
Drug: 1/2 therapeutic dose — 5 volunteers + 1 replacement volunteer will recieve 1/2 therapeutic dose of the study drug (parenteral administration).
  Arms: 1/2 therapeutic dose
Drug: full therapeutic dose — 15 volunteers + 3 replacement volunteers will recieve full therapeutic dose of the study drug (parenteral administration).
  Arms: Patients with a verified diagnosis of COVID-19
Drug: Patients with a verified diagnosis of COVID-19 — 10 volunteers with a verified diagnosis of COVID-19 will recieve full therapeutic dose of the study drug (parenteral administration).
  Arms: full therapeutic dose

SUMMARY:
A two-stage open-label, prospective, safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity study with participation of healthy volunteers in three dose-escalation groups and patients with a confirmed diagnosis of COVID-19.

ELIGIBILITY:
INCLUSION CRITERIA

Stage 1

Each potential volunteer for inclusion in Stage 1 of the Study should meet all of the following criteria:

1. Written Informed Consent to participate in the Study.
2. Men and women, age limits: min.: 18, max.: 45.
3. Healthy according to the results of a medical examination: no history of pathology in the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary, immune and endocrine systems, or blood, which may affect the safety of the volunteer and the assessment of the Study results (no diseases or clinically significant abnormalities were revealed by clinical, instrumental, and laboratory tests).
4. Negative test result for COVID-19, determined by PCR at the screening.
5. No contact with COVID-19 patients for at least 14 days prior to inclusion in the Study (according to information provided by potential volunteer).
6. Negative test result for presence of IgM antibodies to SARS CoV2 by enzyme-linked immunosorbent assay.
7. The result of IgG to S-protein or RBD of no more than x3 IGRI (or no more than 30 BAU) to SARS CoV2 by enzyme-linked immunosorbent assay, regardless of the previous immune status.
8. Consent to the use effective methods of contraception during the entire period of participation in the Study.
9. Body mass index (BMI) is 18.5≤BMI≤30.
10. A negative pregnancy test result based on the results of a urine test (for women of childbearing age).
11. Negative test results for HIV, hepatitis B and C, syphilis.
12. A negative urine test result for presence of narcotic and psychostimulants.
13. A negative alcohol content test.
14. Indicators of general and biochemical blood analysis at screening in the range of 1.1 X VGRI - 0.9 X NGRI.
15. Indicators of immunoglobulin E are not higher than 2 X IGRI.

Stage 2

Each potential volunteer for inclusion in Stage 2 of the Study should meet all of the following criteria:

1. Written Informed Consent to participate in the study.
2. Men and women, age limits: min.: 18, max.: 45.
3. A positive test result for SARS-CoV-2 was obtained < 5 days before the inclusion in the Study, or clinical manifestations began, confirmed later by PCR/rapid test.
4. Oxygen saturation ≥93% without oxygen donation in any way, a diagnosis of COVID-19 is made, provided that symptoms appear no later than 5 days at the time of inclusion in the Study.
5. The presence of several (at least 2) symptoms of mild or moderate severity at the time of inclusion in the Study;
6. At the time of screening, the potential volunteer is not hospitalized due to the severity of the COVID-19 disease;
7. The presence of factors (at least 1) of a high risk of developing severe COVID-19 and / or hospitalization and / or death, according to the Investigator, not limited to the following:

   1. patients not vaccinated against the current strain of the virus
   2. elderly patients (over 60 years of age), including those with additional risk factors
   3. obesity
   4. patients with immunodeficiency, including those taking immunosuppressive drugs for any indication
   5. comorbidities (diabetes mellitus, cardiovascular diseases, coagulopathies, chronic kidney disease, including conditions requiring dialysis, chronic lung diseases, liver diseases, etc.)
8. Consent to the use of effective methods of contraception during the entire period of participation in the Study.
9. The potential volunteer is able to perform visits during the Study.

EXCLUSION CRITERIA

Stage 1

The potential volunteer will not be included in Stage 1 of the Study in the following cases:

1. Inability to read in Russian; inability or unwillingness to understand the essence of the Study. Any other condition that restricts the validity of obtaining informed consent or may affect the volunteer's ability to participate in the Study.
2. Plasma treatment from a recovered COVID-19 patient or MCA against SARS-CoV-2 in the last 3 months.
3. Acute infectious diseases within 2 weeks and non-infectious diseases, exacerbations of chronic diseases within 4 weeks before the screening.
4. The presence of inflammatory or dystrophic changes in the myocardium according to the results of ECG performed on the screening.
5. The volunteer's participation in any other study within the last 90 days.
6. A history of splenectomy.
7. Presence of mental illnesses (registered by psychiatric / mental health facility).
8. Treatment with steroids (excluding hormonal contraceptives) for the last 10 days.
9. Administration of monoclonal antibodies, immunoglobulins or blood products in the last 3 months.
10. Autoimmune diseases or a history of systemic collagenosis that require immunosuppressive therapy.
11. Volunteers who have undergone organ transplants, including bone marrow or peripheral blood stem cell (PSCC) transplants.
12. Immunosuppressive drugs and / or immunomodulators intake for 6 months prior to the start of the Study.
13. Any immunodeficiency (for example, hereditary immunodeficiency, acquired immunodeficiency syndrome [AIDS], etc.,).
14. Pregnancy or breast-feeding.
15. Systolic blood pressure less than 100 mmHg or higher than 139 mmHg; diastolic blood pressure less than 60 mmHg or higher than 90 mmHg; heart rate less than 60 beats / min or more than 100 beats / min.
16. A burdened allergic history (including, but not limited to, major multiform erythema, toxic epidermal necrolysis, angioedema, polymorphic exudative eczema, a history of serum sickness, hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to the components of the drug, etc.).
17. History of severe infusion reactions
18. Diabetes mellitus or other forms of glucose tolerance disorders;
19. The medical history of malignant neoplasms, with the exception of basal cell or squamous cell epithelial skin carcinomas, which were removed without any signs of metastasis for 3 years.
20. Blood donation (450 ml or more of blood or plasma) less than 2 months before the start of the Study;
21. Taking narcotic and psychostimulant drugs at the present time or according to the anamnesis.
22. Drinking alcohol above the low-risk level: no more than 20 grams of pure alcohol per day, no more than 5 days a week, alcohol intake within 48 hours before the study drug administration.
23. Smoking: more than 10 cigarettes a day.
24. Planned hospitalization and / or surgical intervention during the period of participation in the Study, as well as 4 weeks before the expected date of study drug administration.
25. The presence of a concomitant disease that may affect the evaluation of the Study results or that, in the opinion of the Investigator, will not allow the volunteer to participate in the Study or may affect the conduct of the study and/or its results (including the assessment of safety parameters), any conditions that, in the opinion of the Investigator (doctor), may be a contraindication to participation in the Study.
26. The weight of a potential volunteer is less than 45 and more than 100 kg (even if the BMI of the volunteer corresponds to the norm-item 8 of the inclusion criteria).

Stage 2

The potential volunteer will not be included in Stage 2 of the Study in the following cases:

1. Inability to read in Russian; inability or unwillingness to understand the essence of the research. Any other conditions that limit the validity of obtaining informed consent or may affect the patient's ability to participate in the Study.
2. Pregnancy and lactation.
3. Severe and extremely severe course of COVID-19:

   * Blood oxygen saturation at rest according to pulse oximetry (SpO2) < 93% OR
   * PaO2 / FiO2 ≤ 300 mmHg OR
   * Respiratory failure and the need for invasive mechanical ventilation (with tracheal intubation) or ECMO; OR
   * Septic shock OR
   * Multiple organ failure
4. Previous plasma therapy from a recovered patient with COVID-19 or other mAb drugs against SARS CoV-2 for the treatment of COVID-19 disease that is ongoing at the time of inclusion in the Study.
5. The patient is currently hospitalized or, according to the Investigator, may require hospitalization in the next 24 hours due to the severity of the infection.
6. Oxygen therapy is required due to COVID-19 disease or an increase in the baseline oxygen flow rate due to COVID-19 disease is required in individuals on chronic oxygen therapy due to a non-COVID-19 comorbidity.
7. Confirmed active tuberculosis, AIDS (according to medical history, registration).
8. The presence of any life-threatening concomitant disease in a state of decompensation, which, in the opinion of the Investigator, makes the patient unsuitable for inclusion in the Study;
9. Body weight less than 40 kg.
10. Participation in any other study within the last 90 days.
11. Artificial lung ventilation is required or an unavoidable need for mechanical ventilation is predicted in the next 24 hours based on the patient's current condition.
12. A suspected or proven serious active bacterial, fungal, viral, or other infection (other than COVID-19) that the Investigator believes may pose a risk to the patient and affect the assessment of Study endpoints.
13. There are concomitant diseases that require surgical intervention within the next month.
14. A burdened allergic history (including, but not limited to, erythema majora multiforme, toxic epidermal necrolysis, angioedema, polymorphic exudative eczema, a history of serum sickness, hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to the components of the study drug, etc.).
15. A history of severe infusion reactions.
16. Alcohol or drug addiction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | within 28 days after administration of the study drug

IPD SHARING:
Plan to Share IPD: No